CLINICAL TRIAL: NCT05750732
Title: Investigation of the Relationship Between Weight Loss Diet and Circadian Gene CLOCK 3111T/C Polymorphism
Brief Title: Weight Loss and CLOCK 3111T/C Polymorphism
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hande Gül Ulusoy Gezer, Research Assistant, Hacettepe University
Other Study IDs: GO 22/1321
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-10

CONDITIONS: Polymorphism, Restriction Fragment Length; Obesity
Keywords: obesity; circadian rhythm; polymorphism; CLOCK gene; weight loss diet
MeSH Terms: conditions — Obesity | interventions — Diet, Reducing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group: Age range 20-50, BMI range of 25-40 kg/m2
  Interventions: Behavioral: Weight loss diet
- Control group: Age range 20-50, BMI range18.5-24.9 kg/m2

INTERVENTIONS:
Behavioral: Weight loss diet — Participants in the study group will be given training on the weight loss diet, which is a routine part of their treatment.
  Groups: Study group

SUMMARY:
The goal of this observational study is to investigate the relationship of CLOCK 3111T/C (rs1801260) gene variant with nutritional habits, nutritional status, chronotype, sleep quality, some biochemical parameters in overweight or obese individuals and to observe its effect on weight loss diet intervention. The main questions it aims to answer are:

* Is the frequency of carrying the CLOCK 3111T/C (rs1801260) gene risk allele different between individuals with normal body weight and those who are overweight or obese?
* Do those with the CLOCK 3111T/C (rs1801260) risk allele have a higher frequency of evening chronotype and a shorter sleep duration?
* Is the effect of CLOCK 3111T/C (rs1801260) gene alleles different on weight loss diet response in overweight or obese individuals? A questionnaire will be applied to the individuals in both groups (normal body weight and overweight/obese individuals) to evaluate their general characteristics, eating habits, adherence to Mediterranean diet, DASH and MIND. In addition, anthropometric measurements, 3-day food consumption record and 3-day physical activity record will be taken from individuals. CLOCK 3111T/C (rs1801260) gene variant analysis in whole blood, adiponectin and leptin hormones in serum samples will be studied. Participants those who are overweight/obese will be asked to follow a weight loss diet for 3 months.

Researchers will compare participants with normal body weight and those who are overweight or obese to see if there is a difference between the frequency of carrying the CLOCK 3111T/C (rs1801260) gene risk allele.

ELIGIBILITY:
Inclusion Criteria:

* Be in the 20-50 age range
* BMI in the range of 25-40 kg/m2 for the study group
* BMI of 18.5-24.9 kg/m2 for the control group

Exclusion Criteria:

* Those with type 1 diabetes
* Those with Type 2 diabetes who take insulin therapy or use oral diabetes medication
* Those who use drugs for weight loss
* Those with unstable cardiovascular disease
* Those with kidney or liver failure
* Presence of diagnosed malabsorption (celiac disease, Crohn's, ulcerative colitis)
* Those who have undergone bariatric surgery
* Those who are pregnant or breastfeeding
* Menopausal women
* Those who use corticosteroids
* Those with severe endocrine disorders (hypothyroidism, hyperthyroidism, hypopituitarism)
* Those with psychiatric or neurological disease
* Weight change of >5% in the last 6 months
* Those with malignant tumors
* Those with eating disorders
* Shift workers
* Relatives
* People from different ethnic backgrounds

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study consists of overweight or obese individuals who applied to Hacettepe University Adult Hospital Endocrinology outpatient clinic. Individuals will be included in the study after being evaluated by the responsible physician and dietitian in Hacettepe University Adult Hospital Endocrinology outpatient clinic in terms of inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 12 weeks
  Body weight (kg) at 12 weeks minus weight at baseline (kg)
Change in dietary energy and nutrient intakes | Baseline to 12 weeks
  Energy and nutrients intakes will be assessed using a dietary recall method at baseline, 4th week, 8th week and at end of the intervention
Circadian CLOCK gene polymorphism | 1 day
  Comparative analysis of the frequency distributions of genotypes and alleles of 3111T/C CLOCK gene polymorphism will be carried out both in study and control group

SECONDARY OUTCOMES:
Change in sleep quality | Baseline to 12 weeks
  Using 19-item Pittsburg Sleep Quality Index (PSQI)
Change in adherence to Mediterranean diet | Baseline to 12 weeks
  Using the 14-item Mediterranean Diet Adherence Screener (MEDAS)
Change in adherence to DASH | Baseline to 12 weeks
  Using the 11-item Dietary Approaches to Stop Hypertension-Quality (DASH-Q)
Change in adherence to MIND | Baseline to 12 weeks
  Using the 14-item The Mediterranean-DASH Diet Intervention for Neurodegenerative Delay (MIND) score
Change in chronotype | Baseline to 12 weeks
  Using the 19-item The Morningness-Eveningness Questionnaire (MEQ)
Change in eating behaviors | Baseline to 12 weeks
  Using the 18-item The Three-Factor Eating Questionnaire (TFEQ-18)
Change in night eating behaviors | Baseline to 12 weeks
  Using the 16-item The Night Eating Questionnaire (NEQ)
Change in serum adiponectin and leptin level | Baseline to 12 weeks
  Using ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: Hanife Seda Oğuz Baykal, Dr, Study Chair — Hacettepe University; Erdem Karabulut, Prof, Study Chair — Hacettepe University; Neslişah Rakıcıoğlu, Prof, Study Director — Hacettepe University; Hande Gül Ulusoy Gezer, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided